CLINICAL TRIAL: NCT04844229
Title: Bilateral Sphenopalatine Ganglion Block With or Without Bilateral Greater Occipital Nerve Block for Treatment of Obstetric Post-Dural Puncture Headache After Spinal Anesthesia
Brief Title: Bilateral Sphenopalatine Ganglion Block With or Without Bilateral Greater Occipital Nerve Block for Treatment of Obstetric Post-Dural Puncture Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Amr Shaaban Elshafei, Principle Investigator, Zagazig University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6868
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2022-10-18 (Actual); Status verified 2022-10

CONDITIONS: Post-Dural Puncture Headache
MeSH Terms: conditions — Post-Dural Puncture Headache | interventions — spirogermanium; Dental Occlusion

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): 21 patients will receive conservative management for PDPH in the form of oral paracetamol 1000 mg/8hours, and caffeine 300-500 mg/day, 1000 mL 0.9% normal saline infusion over the initial 4 hours with increasing oral fluids and bed rest to be maintained. After 6 hour of starting treatment if the above measures failed to control pain with the VAS ≥ 4 non-steroidal anti-inflammatory drugs (NSAID) will be added in the form of ketorolac 30 mg IV which can be repeated every 12 hours if needed. Participants will be followed up after 1 hour, 6 hours and 24 hours with assessment of VAS score, modified Lybecker clas¬sification score and TCD parameters. EBP will be considered after 24 hours of treatment if pain still not controlled with VAS ≥ 4 and modified Lybecker clas¬sification score ≥ 2 and after patients' consent.
- Interventional group (Active Comparator): 21 patients will receive the same conservative management as in control group together with bilateral transnasal sphenopalatine ganglion block.
  After one hour Participants who will show improvement in pain scores will be followed up after 6 hours and 24 hours, while, patients who will show persistent headache will be subjected for bilateral ultrasound guided greater occipital nerve block.
  then these patients will be assessed after 1 h, 6 h, and 24 h of the block. If still suffering epidural blood patch will be indicated and performed after gaining patients' consent.
  Interventions: Procedure: Bilateral transnasal sphenopalatine ganglion block.; Procedure: Bilateral ultrasound guided greater occipital nerve block.

INTERVENTIONS:
Procedure: Bilateral transnasal sphenopalatine ganglion block. — SPG block will be performed with the patient in supine position using cotton-tipped plastic hollow applicator inserted in the nose with the swab soaked in 1.5 ml 10%lignocaine. The applicator will be inserted parallel to the floor of the nose until resistance encountered. The swab will be rested in the pterygopalatine fossa superior to the middle turbinate and removed after 10 min. This procedure will be repeated in the other nostril too.
  Other Names: (SPG) block.
  Arms: Interventional group
Procedure: Bilateral ultrasound guided greater occipital nerve block. — GONB will be performed with the patients lying in prone position using high frequency (6-13 MHz) probe of Siemens Acuson X300 machine placed in transverse orientation lateral to external occipital protuberance parallel to the superior nuchal line to detect occipital artery where the nerve is located medial to it 1.5inch; then 20 gauge needle will be inserted out of plane to avoid vascular injury. 4 ml of treatment solution containing 2.5 mg/ml bupivacaine and 1 mg/ml dexamethasone (prepared by adding 2 ml bupivacaine 0.5% + 1 ml dexamethasone + 1 ml saline) will be injected on each side.
  Other Names: (GONB).
  Arms: Interventional group

SUMMARY:
Post-dural puncture headache is a common complication, following neuraxial techniques. The obstetric population is particularly prone to PDPH. Therefore, treatment of PDPH is a key issue in obstetric anesthesia. Conservative treatment for PDPH includes adequate hydration, systemic analgesia with paracetamol and non-steroidal anti-inflammatory drugs and increased caffeine intake, as well as bed rest. If these measures are unsuccessful, the gold standard for the treatment of PDPH is the epidural blood patch which is an invasive technique.

The use of nerve blocks for treating headache symptoms are well known techniques that have been previously used for managing some specific types of chronic headache such as cervicogenic headache, cluster headache, migraine, and occipital neuralgia and there are some recently published studies reporting that these blocks may be beneficial in treating PDPH and the available evidence although showing improvements in the visual analogue (VAS) scores and a reduced number of patients requiring an epidural blood patch, but it is still poor.

Less invasive techniques such as SPG block and GONB are attractive therapeutic options which may eliminate the need for EBP in obstetric patients suffering from PDPH. Up to the best of our knowledge this is the first randomized trial to investigate the analgesic efficacy of adding SPG block either alone or in combination with GONB to PDPH treatment.

DETAILED DESCRIPTION:
Post-dural puncture headache (PDPH) is a relatively common complication following dural puncture which is more frequently noted in parturients undergoing cesarean section (CS) under neuraxial anesthesia. The mechanism of nociception in PDPH is still indistinct. However, it is thought to be related to the decrease in intracranial pressure caused by the cerebrospinal fluid (CSF) leak through the dural defect leading to a downward pull of intracranial nociceptive structures which is further exacerbated by compensatory cerebral vasodilation. Managing Post-dural Puncture Headache is a challenge for most anesthesiologists as the gold standard and definitive treatment; epidural blood patch (EBP) itself can lead to inadvertent dural puncture that caused the complication in the first place. Medical and conservative management of PDPH may not provide symptomatic relief and anesthesiologists are on a constant lookout for techniques that can provide immediate and sustained relief from this debilitating complication.

The use of regional techniques and nerve blocks for the treatment of headache symptoms are well known techniques. The transnasal sphenopalatine ganglion (SPG) block which is an easy block that requires minimal training was shown to be helpful in the PDPH treatment with promising results. The SPG surrounded by mucous membrane within the posterior nasal turbinate, is a parasympathetic ganglion of cranial nerve (CN) VII which mediates intracranial vasodilation. The role of this block in PDPH management may be due to the vasoconstriction resulting from the parasympathetic block. Additionally, its relationship to the fifth cranial nerve (trigeminal nerve) may simultaneously relieve the frontal headache.

Another regional technique that can be used is the Greater Occipital Nerve Block (GONB) that has been previously used for managing some specific types of chronic headache such as cervicogenic headache, cluster headache, migraine, and occipital neuralgia and there are some recently published studies reporting that GONB may have a beneficial role in PDPH management. In addition, it is a superficial block which can be done at the patient's bedside under ultrasound guidance. The greater occipital nerve is the main sensory nerve of the occipital region that arises from the dorsal ramus of cervical spinal nerve II. The neuromodulation effect together with decreased central sensitivity resulting from meningial and paraspinal muscles irritation as well as blocking the spinal cord dorsal horn afferent fibers may explain the role of GONB in relieving PDPH symptoms. Moreover, the sensitive neurons of the upper cervical cord are close to the trigeminal caudal nucleus. Therefore, its afferences may also be blocked with this technique.

The available evidence of these blocks for treating PDPH although showing improvements in the visual analogue (VAS) scores and a reduced number of patients requiring an epidural blood patch, but it is still poor. Moreover, there are some clinical scenarios in which the patient may refuse treatment with the epidural blood patch, or there may be a contraindication for its use. Hence, we hypothesized those obstetric patients who are particularly prone to PDPH may get benefit from these less invasive techniques and that these blocks may be added to the treatment of patients suffering from PDPH in order to avoid the invasive EBP.

ELIGIBILITY:
Inclusion Criteria:

* Patient acceptance.
* Age 21- 40 years old.
* Post-partum females suffering PDPH with visual analogue score (VAS) ≥ 4 and modified Lybecker classification score ≥ 2
* ASA II (due to pregnancy).
* Body mass index < 35Kg/m2
* Accepted mental state of the patient.

Exclusion Criteria:

* Emergent cesarean section.
* Hypertensive disorders of the pregnancy.
* History of allergy to local anesthetics.
* History of chronic headache, migraine, convulsions, and cerebrovascular accident.
* Contraindication to spinal anesthesia: coagulopathy, infection at site of injection.
* Inadequate temporal window

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2021-06-20 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
visual analogue scale | 24 hours
  pain score

SECONDARY OUTCOMES:
Trans-Carnial Doppler | 24 hours
  to measure mean flow velocity and the Gosling pulsatility index

CONTACTS AND LOCATIONS:
Overall Officials: Sherif Mo Mowafy, MD, Study Director — Assistant professor of Anesthesia & Surgical Intensive Care Faculty of Medicine - Zagazig University
Locations (1):
- Zagazig University, Zagazig, Sharqia Province, Egypt